CLINICAL TRIAL: NCT02325063
Title: Leukocyte and Platelet Rich Plasma Versus Type A Botulinum Toxin Versus Glucocorticoids for the Treatment of Lateral Epicondylalgia: a Randomized, Multicenter, Double-blind, Therapeutic Trial With Three Parallel Arms
Brief Title: Evaluation of Three Types of Injection for the Treatment of Lateral Epicondylalgia
Acronym: LET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Discontinuation of production of the investigational medicinal product (PRP)
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-I/2013/MV-01; 2014-001300-22 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Epicondylitis, Lateral Humeral; Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PRP-L Group (Experimental): Patients randomized to this group will be treated with an injection of Leukocyte and Platelet Rich Plasma (PRP-L).
  Intervention: PRP-L Injection
  Interventions: Drug: PRP-L Injection
- Botox Group (Active Comparator): Patients randomized to this group will be treated with an injection of Type A Botulinum Toxin (Xeomin®, MERZ).
  Intervention: Botox injection
  Interventions: Drug: Botox injection
- Corticoid Group (Active Comparator): Patients randomized to this group will be treated with an injection of Corticoids.
  Intervention: Corticoid injection
  Interventions: Drug: Corticoid injection

INTERVENTIONS:
Drug: PRP-L Injection — Patients will be treated with an injection of leukocyte and platelet rich plasma.
  Arms: PRP-L Group
Drug: Botox injection — Patients will be treated with an injection of Type A Botulinum toxin.
  Other Names: Type A Botulinum toxin injection; Xeomin®, MERZ
  Arms: Botox Group
Drug: Corticoid injection — Patients will be treated with an injection of Corticoids.
  Arms: Corticoid Group

SUMMARY:
The primary objective of this study is to compare the evolution of pain profiles among patients suffering from lateral epicondyalgia (tennis elbow) following three types of treatment: PRP-L injection versus type A botulinum toxin injection versus corticoid injection.

DETAILED DESCRIPTION:
The secondary objectives are to compare the following among the three groups:

A- The global efficacy of each treatment defined by a minimum reduction of 25% in average pain over the last 24 hours between 0 and 6 months.

B- The evolution of average pain over the last 24 hours between 0 and each different time frame (3 weeks, 6 weeks, 3 months and 6 months).

C- The evolution of maximum pain scores using nocturnal post-effort (Jamar grip test) visual analog scales (VAS) between day 0, 3 weeks, 6 weeks, 3 months and 6 months.

D- The perception of change on the Patient's Global Impression of Change score (PGIC) at 3 and 6 months E- The evolution of PRTEE scores at 0, 3 and 6 months F- Adverse events at 3 weeks, 6 weeks, 3 months and 6 months. G - Quality of life and utility via the SF-12 at 3 and 6 months. H- The consumption of analgesics.

ELIGIBILITY:
General inclusion criteria:

* The patient must have given free and informed consent and signed the consent
* The patient must be affiliated or beneficiary to a health insurance plan
* The patient is available for 6 months of follow-up
* Woman of childbearing age using contraception

Inclusion criteria for the target population: the patient has a side epicondylalgia objectified by:

* Clinical criteria: symptoms lasting for more than 6 weeks and less than 12 months. The list of symptoms to be present are: pain on palpation of the lateral epicondyle, pain in the lateral epicondyle during blocked contraction
* Therapeutic: less than two injections of corticosteroids performed, and the last such injection was performed at least 3 months before inclusion

General non-inclusion criteria:

* The patient is participating in another study
* The patient is exclusion period determined by a previous study
* The patient is under judicial protection
* The patient is under guardianship or curatorship
* The patient refuses to sign the consent
* Woman of childbearing age not using contraception
* Impossible to correction inform the patient about the study

Non-inclusion criteria for investigational and auxiliary medicinal products:

* The patient has at least one of the contra-indications listed in the SPC for Xeomin and ALTIM:
* Hypersensitivity to Botulinum neurotoxin type A or Cortivazol
* Hypersensitivity to any of the excipients used in the composition of XEOMIN (Human albumin, sucrose) and / or ALTIM (Benzyl alcohol, carmellose sodium, sodium chloride, cetylpyridinium chloride, polysorbate 80)
* Generalized disorders of muscle activity (eg myasthenia gravis, Lambert-Eaton syndrome).
* Severe coagulation disorders, anticoagulation in progress (ticlopidine, clopidogrel, other antiplatelet or antithrombotic agents)
* Presence of a local or general infection, suspected infection, infection at the proposed injection site.

Non-inclusion criteria for the medical device used for the PRP samples (SmartPReP2 sampling system):

* Clinical or laboratory evidence for sepsis
* Taking aspirin or other drugs altering platelet function in the previous 3 days
* Patient with the platelet dysfunction disorders

Non-inclusion criteria for interfering diseases or conditions:

* The patient is pregnant, parturient or she is breastfeeding
* The patient has an allergy to botulinum toxin type A and / or glucocorticoids
* The patient has medial epicondylalgia
* The patient has a history of elbow surgery
* The patient has any of the following conditions: immunodeficiency, rheumatic disease, hepatitis, diabetes, another disease of the ipsilateral limb, neurological disorder (radiculopathy, compression of the radial nerve), any myopathy (all etiologies)
* The patient received treatment with corticosteroids in the last 3 months
* The patient is being treated with long-term anti-platelet medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) for pain over the last 24 hours | 6 months versus Baseline (day 0)
  score varying from 0 to 10

SECONDARY OUTCOMES:
Visual analog scale for pain over the last 24 hours | Baseline (day 0)
  score varying from 0 to 10
Visual analog scale for pain over the last 24 hours | 3 weeks
  score varying from 0 to 10
Visual analog scale for pain over the last 24 hours | 6 weeks
  score varying from 0 to 10
Visual analog scale for pain over the last 24 hours | 3 months
  score varying from 0 to 10

OTHER OUTCOMES:
Global efficacy | 6 months
  Defined as the proportion of patients for whom a decrease in visual analog scales for pain over the last 24 hours of at least 25% has been observed over the past 6 months.
VAS for pain after a Jamar grip test | Baseline (day 0)
  score varying from 0 to 10
VAS for pain after a Jamar grip test | 3 months
  score varying from 0 to 10
VAS for pain after a Jamar grip test | 6 months
  score varying from 0 to 10
PRTEE Score | Baseline (day 0)
  The Patient-Rated Tennis Elbow Evaluation
PRTEE Score | 3 months
  The Patient-Rated Tennis Elbow Evaluation
PRTEE Score | 6 months
  The Patient-Rated Tennis Elbow Evaluation
Patient Global Impression of Change | 3 months
  score varying from 1 to 7
Patient Global Impression of Change | 6 months
  score varying from 1 to 7
Number of patients with adverse effects | Baseline (day 0)
Number of patients with adverse effects | 3 weeks
Number of patients with adverse effects | 6 weeks
Number of patients with adverse effects | 3 months
Number of patients with adverse effects | 6 months
The SF 12 questionnaire | 3 months
The SF 12 questionnaire | 6 months
The consumption of analgesics. | Baseline (day 0)
The consumption of analgesics. | 3 weeks
The consumption of analgesics. | 6 weeks
The consumption of analgesics. | 3 months
The consumption of analgesics. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Vaucher, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes